CLINICAL TRIAL: NCT00301353
Title: Effects of Phytoestrogen-rich Diets on Bone Turnover in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: European Commission (Other); National Institute for Research on Food and Nutrition (Unknown); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Phytos QLRT-2000-00431-WP3
Record Dates: First submitted 2006-03-03; First posted 2006-03-10 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2002-10

CONDITIONS: Osteoporosis
Keywords: early menopause; isoflavones/phyto-estrogens; bone metabolism; bone mineral density; hormones
MeSH Terms: conditions — Osteoporosis; Primary Ovarian Insufficiency

INTERVENTIONS:
Drug: Isoflavones-enriched foods

SUMMARY:
Osteoporosis is a major health problem. It was hypothesized that isoflavone-containing products may be a potential alternative to HRT for preventing bone loss during the menopausal transition. We investigated whether one-year consumption of isoflavone-enriched foods affected bone mineral density, bone metabolism and hormonal status in early postmenopausal women in a randomized double-blind, placebo controlled parallel multi-centre trial.

DETAILED DESCRIPTION:
Two hundred and thirty-seven healthy early post-menopausal women (age 53 ± 3 y; time since last menses 33 ± 15 months) consumed isoflavone-enriched foods providing a mean daily intake of 110 mg isoflavone aglycones or control products for 1 yr whilst continuing their habitual diet and lifestyle. Outcome measures included bone mineral density of lumbar spine and total body, markers for bone formation and bone resorption, hormones, isoflavones in plasma and urine, safety parameters and reporting of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the:

   * health and lifestyle questionnaire
   * physical examination
   * results of the pre-study laboratory tests
2. Caucasian women
3. Postmenopausal (≥12 - ≤60 months since last menses), determined by

   * interview
   * FSH level ≥ 20 IU/l
4. Body Mass Index (BMI) ≥22 - ≤29 kg/m2
5. Voluntary participation
6. Having given their written informed consent
7. Willing to comply with the study procedures
8. Willing to accept use of all nameless data, including publication and the confidential use and storage of all data
9. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

1. Participation in any clinical trial including blood sampling and/or administration of products up to 90 days before Day 01 of this study
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalatory administration of products
3. Osteoporosis, determined by

   * Questionnaire (spontaneous bone fractures, use of medication to treat osteoporosis)
   * DXA scans of the lumbar spine between day -14 and day 1 of the study; exclusion threshold is set at -2z score of BMD
4. Severe scoliosis (curvature of the spine) that could interfere with the ability of the subject to go through the DXA scanning procedure and/or with a correct reading of the DXA scans
5. Having a history of medical or surgical events that may significantly affect the study outcome, including:

   * surgical menopause (including hysterectomy)
   * antecedents and high familiar incidence of breast and/or endometrial cancer
   * gastrointestinal disease (Crohn's, short bowel syndrome, coeliac disease, gastroenteritis episodes the month before the start of the study)
   * hepatic disease (acute or viral hepatitis, chronic hepatitis)
   * cardiovascular disease and thrombosis
   * impaired renal function
   * severe immune disease
   * endocrine diseases (hyperthyroidism, hyperparathyroidism, IDDM, NIDDM)
6. Food allergy as reported by the subject (with special emphasis on soy products) and reported allergy for sunscreen products
7. Use of concomitant medication including

   * Hormonal replacement therapy (during the study and within the last 6 months before day 01 of the study)
   * Current use of corticosteroids (including Aerosol therapy) or past use for more than 10 days within the last 6 months
   * Osteoporosis treatment (biphosphonates, SERM's, calcitonin, injectable PTH)
   * Other medications known to affect bone metabolism (statins). Use of antibiotics will be carefully recorded.
8. Change in smoking habits for the last 2 months
9. Alcohol consumption > 21 units (drinks)/week
10. Reported unexplained weight loss or gain of > 5 % of usual body weight in the month prior to the pre-study screening
11. Reported slimming or medically prescribed diet
12. Professional sportswomen (> 10 hours extensive sports/week)
13. Reported vegan, vegetarian, macrobiotic food intake
14. Regular intake of soy based foods (>2 servings per week). Participation is possible when the subject is prepared to stop consumption from screening until the end of the study
15. Taking supplements containing isoflavones, in the 3 months prior to enrolment and during the study. Subjects should not start taking calcium and vitamin D supplements during the study. However, subjects who already take calcium and vitamin D supplements should maintain this intake during the study
16. Recent blood or plasma donation (<1 month prior to the start of the study)
17. Not willing to stop blood or plasma donation during the study
18. TNO Nutrition and Food Research personnel, their partner and their first and second generation relatives
19. Not having a general practitioner
20. Not willing to accept information-transfer concerning participation in the study, or information regarding his/her health. For example, laboratory results, findings at health and lifestyle questionnaire interview, or physical examination and eventual adverse events communicated to and from their general practitioner
21. Mental status incompatible with the proper conduct of the study

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-10; Study Completion 2004-07

PRIMARY OUTCOMES:
Bone mineral density of total body and lumbar spine (DXA)

SECONDARY OUTCOMES:
Blood and urine markers for bone formation (ALP, PINP) and bone resorption (DPD, PYD)
Hormones (estradiol, FSH, LH, SHBG)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Brink, PhD, Principal Investigator — TNO
Locations (3):
- Institute National de la Recherche Agronomique, Saint-Genès-Champanelle, France
- National Institute for Research on Food an Nutrition, Rome, Italy
- TNO Quality of Life, Zeist, Netherlands

REFERENCES:
- [Derived] Brink E, Coxam V, Robins S, Wahala K, Cassidy A, Branca F; PHYTOS Investigators. Long-term consumption of isoflavone-enriched foods does not affect bone mineral density, bone metabolism, or hormonal status in early postmenopausal women: a randomized, double-blind, placebo controlled study. Am J Clin Nutr. 2008 Mar;87(3):761-70. doi: 10.1093/ajcn/87.3.761. PMID 18326616